CLINICAL TRIAL: NCT00807183
Title: Indoor Woodsmoke PM and Asthma: a Randomized Trial
Brief Title: Indoor Woodsmoke PM and Asthma
Acronym: ARTIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Anthony J. Ward, Associate Professor, National Institute of Environmental Health Sciences (NIEHS)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16336-CP-001
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tx1 (Placebo Comparator): Inactive air filter
  Interventions: Other: inactive air filter
- Tx2 (Experimental): New EPA-certified woodstove
  Interventions: Other: woodstove
- Tx3 (Experimental): Active air filter
  Interventions: Other: Active air filter

INTERVENTIONS:
Other: woodstove — installation of new EPA-certified woodstove
  Arms: Tx2
Other: inactive air filter — air filter units without filter in place
  Arms: Tx1
Other: Active air filter — air filter units correctly operating
  Arms: Tx3

SUMMARY:
Although particulate matter (PM) exposures have been linked with poor respiratory health outcomes, most of these studies have focused on airsheds with urban and industrial sources of PM2.5. Woodsmoke-derived PM also contributes to ambient PM in these urban areas, and is the major source of PM in many US rural or peri-urban areas, as well as in many communities within developing countries. This study will focus on indoor air quality and clinically relevant changes in health effects among asthmatics living in homes whose primary heating sources are non EPA-certified woodstoves. The Primary Aim of this study is to assess the efficacy of residential interventions to reduce indoor PM exposure from woodstoves and the corresponding improvements in quality of life and health outcomes for asthmatic children. The study area for this project will be three rural communities in western Montana and Idaho, including one Indian Reservation. This study will use a three arm (Tx1, Tx2, and Tx3) randomized placebo-controlled intervention trial. The interventions will be at the household level, and exposure and outcomes will be assessed for one asthmatic child in each household. Households in Tx1 will receive inactive high efficiency particulate air (HEPA) devices and will serve as the placebo group. Households in Tx2 will receive a new EPA-certified woodstove, while households in Tx3 will receive active HEPA devices. The Secondary Aims of this study are to assess the impact of these interventions on residential PM2.5 exposures and other health outcomes. Secondary exposure outcomes measured prior to and following the intervention will include PM2.5 mass, chemical woodsmoke markers on PM2.5 filters (including levoglucosan and abietic acids), and biomarkers of woodsmoke exposure. Secondary asthma-related health outcomes measured prior to and following the intervention will include peak expiratory flow (PEF) and forced expiratory volume in first second (FEV1), biomarkers in exhaled breath condensate, and frequency of asthma symptoms, medication usage, and healthcare utilization. To our knowledge, this will be the first randomized trial in the US to utilize a woodsmoke intervention to assess the impact of the consequent reductions in indoor PM on health outcomes in a susceptible population. The results from this project will be translatable to other regions in the US and the world where biomass burning is commonly used for heating and cooking.

DETAILED DESCRIPTION:
SPECIFIC AIMS Although particulate matter (PM) exposures have been linked with poor respiratory health outcomes, most of these studies have focused on populated airsheds with urban and industrial sources of PM2.5. In less-urban areas, residential woodstoves are not only major sources of ambient PM2.5, but can result in significant woodsmoke exposures in the indoor environment. This study will focus on indoor air quality and associated health effects among asthmatic children living in homes whose primary heating sources are non EPA-certified woodstoves. The primary aim of this study is to assess the efficacy of residential interventions to reduce indoor PM exposure from woodstoves and the corresponding improvements in quality of life and health outcomes for asthmatic children. This study will allow us to characterize the woodsmoke effects on asthmatic conditions and evaluate clinically meaningful health outcomes among asthmatics. This will be the first randomized controlled trial in the US to utilize a woodsmoke-targeted intervention and assess the impact of the consequent reductions in indoor PM on health outcomes in a susceptible population. The results from this project will be translatable to other regions in the US and the world where biomass burning is commonly used for heating or cooking.

This study will use a three arm (Tx1, Tx2, and Tx3) randomized placebo-controlled intervention trial. The interventions will be at the household level, and exposure and outcomes will be assessed for one asthmatic child in each household. Households in Tx1 will receive inactive high efficiency particulate air (HEPA) devices and will serve as the placebo group. One intervention that will be tested in this trial will be the replacement of old woodstoves with cleaner burning EPA-certified woodstoves (Tx2). The other intervention that will be tested will be the installation of HEPA filtration devices within the home (Tx3). Our preliminary data have demonstrated significant reductions in indoor PM using these interventions.

The Primary Aim of this study is to assess the impact on quality of life among asthmatic children following interventions that reduce in-home woodsmoke PM exposures. We will address the following primary hypotheses:

1a. Asthmatic children in homes receiving new woodstoves in Tx2 will have improved asthma-specific quality of life measures compared to asthmatic children in placebo households, Tx1.

1. b. Asthmatic children in homes receiving HEPA filtration units in Tx3 will have improved asthma-specific quality of life measures compared to asthmatic children in placebo households, Tx1.

   The Secondary Aims of this study are to assess the impact of these interventions on residential PM2.5 exposures and other health outcomes. We will address the following secondary hypotheses:
2. a. Changes in winter period PM2.5 exposure in homes receiving interventions (Tx2 and Tx3) will be greater than changes in winter period PM2.5 exposure in placebo households (Tx1). Each treatment group will be evaluated independently against the placebo group. Secondary residential exposure outcomes measured repeatedly during pre- and post-intervention winter periods will include:

   1. PM2.5 mass
   2. chemical woodsmoke markers on PM2.5 filters (i.e., levoglucosan and abietic acids)
   3. biomarkers of woodsmoke exposure in urine and exhaled breath condensate (i.e., levoglucosan and abietic acids)

2b. Changes in winter period health outcomes among asthmatic children living in homes receiving interventions (Tx2 and Tx3) will be more improved than changes in winter period health outcomes in placebo households (Tx1). Each treatment group will be evaluated independently against the placebo group. Secondary exposure outcomes will include:

1. peak expiratory flow (PEF) and forced expiratory volume in first second (FEV1)
2. biomarkers in exhaled breath condensate (i.e., pH and nitric oxide)
3. frequency of asthma symptoms
4. frequency of rescue medication usage
5. healthcare utilization

ELIGIBILITY:
Inclusion Criteria:

* children with moderate to severe asthma living in homes with non EPA-certified woodstove used for heating.

Exclusion Criteria:

-

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2008-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Curtis W Noonan, Ph.D., Principal Investigator — University of Montana; Tony Ward, Ph.D., Principal Investigator — University of Montana
Locations (1):
- University of Montana, Missoula, Montana, United States

REFERENCES:
- [Derived] Noonan CW, Semmens EO, Smith P, Harrar SW, Montrose L, Weiler E, McNamara M, Ward TJ. Randomized Trial of Interventions to Improve Childhood Asthma in Homes with Wood-burning Stoves. Environ Health Perspect. 2017 Sep 13;125(9):097010. doi: 10.1289/EHP849. PMID 28935614
- [Derived] Montrose L, Ward TJ, Semmens EO, Cho YH, Brown B, Noonan CW. Dietary intake is associated with respiratory health outcomes and DNA methylation in children with asthma. Allergy Asthma Clin Immunol. 2017 Feb 27;13:12. doi: 10.1186/s13223-017-0187-8. eCollection 2017. PMID 28261276
- [Derived] Noonan CW, Ward TJ. Asthma randomized trial of indoor wood smoke (ARTIS): rationale and methods. Contemp Clin Trials. 2012 Sep;33(5):1080-7. doi: 10.1016/j.cct.2012.06.006. Epub 2012 Jun 23. PMID 22735495